CLINICAL TRIAL: NCT04456816
Title: An Exploratory, Randomized, Double-blind, Multicenter, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of AP1189 Versus Placebo Administered for 12 Weeks as an add-on to Patients, in ACE Inhibitor or Angiotensin II Receptor Blocker Treatment, With Idiopathic Membranous Nephropathy and Severe Proteinuria
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Treatment With AP1189 in Patients With iMN and Severe Proteinuria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SynAct Pharma Aps (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SynAct-CS003
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Nephrotic Syndrome Due to Idiopathic Membranous Nephropathy; Severe Proteinuria Due to Idiopathic Membranous Nephropathy
MeSH Terms: interventions — N-(3-(1-(2-nitrophenyl)-1H-pyrrol-2-yl)allylidenamino)guanidine

STUDY DESIGN:
Intervention Model Description: Exploratory, randomized, double-blind, multi-center, placebo-controlled 12-weeks study with repeated doses of AP1189
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 mg AP1189 (Experimental): 100 mg AP1189. The treatment is a 12-weeks treatment. Each daily dose will be administered as a tablet
  Interventions: Drug: 100 mg AP1189
- Placebo (Experimental): Placebo. The treatment is a 12-weeks treatment. Each daily dose will be administered as a tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100 mg AP1189 — 100 mg AP1189 tablet
  Arms: 100 mg AP1189
Drug: Placebo — Matching placebo tablet
  Arms: Placebo

SUMMARY:
This study is an exploratory, randomized, double-blind, multicenter, placebo-controlled study with repeated doses of AP1189. The study population will consist of patients with idiopathic membranous nephropathy (iMN) and severe proteinuria who are on ACE inhibitor or angiotensin II receptor blocker treatment.

DETAILED DESCRIPTION:
This study is an exploratory, randomized, double-blind, multicenter, placebo-controlled study with repeated doses of AP1189. The study population will consist of patients with idiopathic membranous nephropathy (iMN) and severe proteinuria who are on ACE inhibitor or angiotensin II receptor blocker treatment.

Following a successful screening, subjects who fulfill the enrollment criteria will be randomized in a 2:1 ratio in group A and B:

* Group A (12 subjects): AP1189 dose 100 mg, once daily for 12 weeks (28 days) as an add-on to any ongoing treatment, including ACE inhibitors/ angiotensin II receptor blocker
* Group B (6 subjects): placebo for 12 weeks (28 days) as an add-on to any ongoing treatment including ACE inhibitors/ angiotensin II receptor blocker.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained prior to initiating any study-specific procedures
* Male and female subjects, 18 to 85 years of age diagnosed with iMN within 6 months prior to inclusion
* Diagnosed as anti-PLA2-Receptor positive by local laboratory within 6 months prior to inclusion
* Severe proteinuria defined by a U-protein/creatinine ratio >3.0 g/g and/or U-albumin/creatinine ratio >2.0 g/g and a P-albumin below the lower normal limit
* eGFR > 30 ml/min/1.73m2
* Treated with ACE- inhibitors or angiotensin II receptor blocker for a minimum of 1 months with a stable systemic arterial blood pressure OR treatment with ACE inhibitors and/or angiotensin receptor blocker was excluded or discontinued due to hypotension, intolerance or other side effect

Only Denmark and Norway:

* Females of child-bearing potential using reliable means of contraception or are post-menopausal
* Females of childbearing potential with negative pregnancy test at screening and baseline

Only Sweden:

* Post-menopausal women or women who are surgically sterilized.

Exclusion Criteria:

* Participation in any other study involving investigational drug(s) during the study and within 4 weeks prior to study entry
* Clinicial findings that in the opinion of the investigator would suggest condition(s) other than iMN as a major cause of severe proteinuria
* Major surgery within 8 weeks prior to screening or planned surgery within 1 month following randomization
* Blood pressure with systolic pressure above 160 mmHg and/or diastolic pressure above 100 mmHg despite antihypertensive treatment will in all cases be considered "uncontrolled"
* Treated with systemic corticosteroids, or other immune suppressive, or immune modulating compounds within 4 weeks prior to screening and during the entire treatment period and until the final visit
* Treated with rituximab within 12 months of screening
* Evidence of active malignant disease
* Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disease
* Pregnant women or nursing mothers
* History of alcohol, drug, or chemical abuse within the 6 months prior to screening
* Any condition that in the view of the investigator would suggest that the patient is unable to comply with study protocol and procedures

Only Sweden:

* Females of child-bearing potential.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Week 12
  Evaluation of Adverse Event
Serious Adverse Events | Week 12
  Evaluation of Serious Adverse Events
ALAT change in plasma samples | Week 12
  Evaluation of ALAT compared with baseline
ASAT change in plasma samples | Week 12
  Evaluation of ASAT compared with baseline
Total bilirubin change in plasma samples | Week 12
  Evaluation of total bilirubin compared with baseline
Alkaline phosphatase change in plasma samples | Week 12
  Evaluation of alkaline phosphatase compared with baseline
Protein change in 24 hours urinary protein excretion | Week 12
  Change of protein in urine excretion compared to baseline measured in 24 h urinary protein excretion

SECONDARY OUTCOMES:
Albumin change in 24 hours urinary protein excretion | Week 12
  Change of albumin in urine excretion compared to baseline measured in 24 h urinary protein excretion

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Birn, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus Universitetshospital, Aarhus, Denmark